CLINICAL TRIAL: NCT03388125
Title: Endoscopic Injection Sclerotherapy Versus N-butyl-2-cyanoacrylate Injection in the Management of Actively Bleeding Esophageal Varices
Brief Title: Endoscopic Injection Sclerotherapy Versus N-butyl-2-cyanoacrylate Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Active bleeding
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Bleeding Esophageal Varices
MeSH Terms: interventions — ethanolamine oleate; Enbucrilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection Sclerotherapy (Active Comparator): 5% ethano lamine oleate
  Interventions: Drug: Injection Sclerotherapy
- N-butyl-2-cyanoacrylate (Active Comparator): N-butyl-2-cyanoacrylate injection group
  Interventions: Drug: N-butyl-2-cyanoacrylate

INTERVENTIONS:
Drug: Injection Sclerotherapy — 5% ethanolamine oleate group
  Other Names: 5% ethanolamine oleate
  Arms: Injection Sclerotherapy
Drug: N-butyl-2-cyanoacrylate — N-butyl-2-cyanoacrylate injection group
  Arms: N-butyl-2-cyanoacrylate

SUMMARY:
Endoscopic Injection Sclerotherapy vs N-butyl-2-cyanoacrylate Injection

DETAILED DESCRIPTION:
Endoscopic Injection Sclerotherapy versus N-butyl-2-cyanoacrylate Injection in the Management of Actively Bleeding Esophageal Varices

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients presented with actively bleeding

Exclusion Criteria:

* other sources of UGIB than esophageal varices, hepatic encephalopathy or hepatocellular carcinoma (HCC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with controlled bleeding | 6 months
  The Number of patients with controlled bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alsebaey, MD, Principal Investigator — Gastroenterology; Mohamed Abdelraouf, MD, Study Director — Gastroenterology; Sherief Abd-Elsalam, MD, Study Director — Hepatology and Gastroenterology
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elsebaey MA, Tawfik MA, Ezzat S, Selim A, Elashry H, Abd-Elsalam S. Endoscopic injection sclerotherapy versus N-Butyl-2 Cyanoacrylate injection in the management of actively bleeding esophageal varices: a randomized controlled trial. BMC Gastroenterol. 2019 Feb 4;19(1):23. doi: 10.1186/s12876-019-0940-1. PMID 30717684